CLINICAL TRIAL: NCT07188675
Title: Effects of Functional Inspiratory Muscle Training on Pulmonary Function, Muscle Thickness, and Core Performance in Patients With Bronchiectasis
Brief Title: Functional Inspiratory Training in Bronchiectasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Kabasakal (Other)
Responsible Party: Sponsor-Investigator, Elif Kabasakal, LECTURER, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISU-2025-005
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Bronchiectasis; Functional Inspiratory Muscle Training
Keywords: bronchiectasis; functional inspiratory muscle training; core stability; muscle thickness; respiratory function
MeSH Terms: conditions — Bronchiectasis; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Inspiratory Muscle Training (FIMT) Group (Experimental): Participants will perform 4 weeks of inspiratory muscle training (IMT) at 50% of maximal inspiratory pressure (MIP), followed by 4 weeks of functional inspiratory muscle training (FIMT) with POWERbreathe. Training includes weekly face-to-face or supervised online sessions and additional unsupervised practice.
  Interventions: Other: Functional Inspiratory Muscle Training (FIMT)
- Inspiratory Mucle Training (IMT) Group (Active Comparator): Participants will perform daily inspiratory muscle training (IMT) for 8 weeks using the POWERbreathe Classic Light Resistance device. Training includes weekly face-to-face sessions with MIP-based load adjustments, plus home practice monitored via WhatsApp.
  Interventions: Other: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training (FIMT) — Participants will begin with Inspiratory Muscle Training (IMT) at 50% of maximal inspiratory pressure (MIP) for 4 weeks. Training will be performed once a week face-to-face, while adherence will be monitored on other days via WhatsApp. During each face-to-face session, MIP will be reassessed and training loads adjusted. Participants will perform 30 dynamic inspiratory efforts twice daily. In the following 4 weeks, Functional Inspiratory Muscle Training (FIMT) will be applied: once face-to-face, twice online under physiotherapist supervision, and twice unsupervised IMT. FIMT exercises will be performed with the POWERbreathe Classic Light Resistance device, consisting of 10 breaths lasting 15-30 seconds in 2 sets. Each session will include warm-up (diaphragmatic breathing and trunk stretches), loading (core stabilization exercises), and cool-down (trunk stretches). IMT intensity will be adjusted weekly using MIP measurement
  Arms: Functional Inspiratory Muscle Training (FIMT) Group
Other: Inspiratory Muscle Training (IMT) — Participants will perform IMT daily for 8 weeks. Training will be conducted once a week face-to-face, while on other days adherence will be monitored via WhatsApp. The group will complete 30 dynamic inspiratory efforts twice daily. The POWERbreathe Classic Light Resistance device (PowerBreathe, IMT Technologies Ltd, Birmingham, UK) will be used to strengthen the diaphragm and chest wall muscles by breathing against a set pressure load. Training intensity will be set at 50% of maximal inspiratory pressure (MIP). After 10-15 consecutive breaths, participants will perform 3-4 recovery breaths before continuing. IMT intensity will be re-adjusted weekly during face-to-face sessions using MIP measurements to maintain 50% loading.
  Arms: Inspiratory Mucle Training (IMT) Group

SUMMARY:
Bronchiectasis is a chronic respiratory disease clinically characterized by recurrent pulmonary exacerbations, chronic cough, and sputum production, and is associated with an increase in the airway-artery ratio and permanent airway dilatation. It is recognized as the third most common chronic respiratory disease after chronic obstructive pulmonary disease (COPD) and asthma. In the International Classification of Diseases and Related Health Problems (ICD-10), it has its own diagnostic code (J47.9).

In bronchiectasis, mucociliary clearance is impaired due to bronchial dilatation, and the insufficient clearance of bacteria and mucus from the respiratory tract leads to persistent infection, inflammation, and further airway damage. Progressive airway damage results in impaired lung function, worsening of symptoms, and, ultimately, respiratory failure and death. It can represent the final pathway of various infectious, allergic, inflammatory, genetic, and degenerative disorders, making it one of the most complex and heterogeneous syndromes. Some patients present with daily symptoms, while others remain asymptomatic except during exacerbations. The most common symptom is chronic cough caused by purulent or mucopurulent sputum. Other symptoms include dyspnea, pleuritic chest pain, wheezing, fatigue, and weight loss. Fever, however, is not a common finding and differs from pneumonia.

The most frequently used classification system categorizes bronchiectasis into varicose, cylindrical, and saccular (cystic) types. In the most severe form, the saccular type, the bronchi lose their structural integrity completely, forming cystic structures filled with secretions. The mildest form is cylindrical, in which the bronchi have thick, straight walls. In the varicose type, localized narrowings are observed. Diagnosis is made following history and physical examination, with high-resolution computed tomography (HRCT) being the most sensitive and specific method, along with sputum culture and chest radiography.

The goals of bronchiectasis treatment are to manage symptoms, prevent complications, and improve quality of life. Both pharmacological and patient-managed interventions are commonly applied. Pharmacological treatments include antibiotics, bronchodilators, and corticosteroids, which are generally administered via inhalation. Patient-managed interventions require active participation and behavioral modification. Within published guidelines, airway clearance techniques are widely described under pulmonary rehabilitation (PR), but there is no consensus regarding PR itself. For individuals with reduced exercise tolerance, participation in PR and engagement in physical activity are recommended. However, research has shown that referral rates to PR are often low, and exercise and physical activity are not consistently prescribed.

Within PR, techniques such as the active cycle of breathing techniques (ACBT), postural drainage, thoracic expansion exercises, and various airway clearance methods are applied, with inspiratory muscle training (IMT) forming an important component. Functional inspiratory muscle training (FIMT) is an IMT program developed by considering not only the ventilatory roles of the respiratory muscles but also their non-respiratory functions. FIMT integrates inspiratory muscle training with core stabilization and postural control exercises. The rhythmic co-contractions of the muscles in the core region support trunk stability and provide the basis for movement. In the first stage of the program, participants receive IMT, and subsequently, core stabilization training and dynamic trunk activation exercises are incorporated into the intervention.

A review of the literature reveals that no studies have investigated the effectiveness of FIMT in adults with bronchiectasis. In our study, we aim to evaluate the effects of FIMT, applied in addition to home-based chest physiotherapy, on pulmonary function, diaphragm thickness, balance, core stability, functional capacity, physical activity, posture, and quality of life in adults with bronchiectasis. Furthermore, we aim to compare these outcomes with those of IMT applied alongside home-based chest physiotherapy. We believe that this approach will contribute to the development of treatment strategies in clinical practice and help address existing gaps in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* Diagnosed with bronchiectasis
* Clinically stable
* Able to cooperate
* Able to walk independently
* Volunteering to participate in the study

Exclusion Criteria:

* History of acute exacerbation and/or hospitalization within the past 4 weeks
* Change in medical treatment within the past month
* Known diagnosed conditions affecting balance (visual, auditory, vestibular, or musculoskeletal disorders)
* Participation in a supervised physiotherapy rehabilitation program within the past 6 months
* History of lung or liver transplantation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) | At baseline (before the intervention) and at the end of the 8th week of intervention
  FEV1 will be assessed using a spirometer (Cosmed Pony FX) under ATS/ERS standards. The measurement will be recorded in liters and as a percentage of the predicted normal value.
Forced Vital Capacity (FVC) | At baseline (before the intervention) and at the end of the 8th week of intervention
  Forced Vital Capacity (FVC) will be measured using a portable spirometer (Cosmed Pony FX, Italy) following ATS/ERS guidelines. Results will be recorded in liters and as a percentage of the predicted value.
FEV1/FVC Ratio | At baseline (before the intervention) and at the end of the 8th week of intervention
  The ratio of FEV1 to FVC (FEV1/FVC) will be calculated to assess airway obstruction. The values will be expressed as a percentage. All procedures will be carried out with standardized spirometry protocols (ATS/ERS) using single-use mouthpieces and filters.
Peak Expiratory Flow (PEF) | At baseline (before the intervention) and at the end of the 8th week of intervention
  PEF will be measured as part of the pulmonary function test using a spirometer. Values will be expressed in liters per second (L/s) and as a percentage of the predicted value. Infection control procedures will include the use of disposable mouthpieces and filters as per device guidelines.
Forced Expiratory Flow (FEF25-75%) | At baseline (before the intervention) and at the end of the 8th week of intervention.
  Forced Expiratory Flow between 25% and 75% of the forced vital capacity (FEF25-75%) will be measured using a portable spirometer (Cosmed Pony FX, Italy) according to ATS/ERS guidelines. Results will be recorded in liters per second and as a percentage of the predicted value.
Maximal Inspiratory Pressure (MIP) | Baseline and Week 8(Post-Intervention)
  Maximal Inspiratory Pressure (MIP) will be measured using a portable electronic mouth pressure device (Micro Medical Micro RPM, UK). The measurement will be performed during maximal inspiratory effort against an occluded airway after full expiration and held for 1-3 seconds. Three trials will be conducted, and the highest value will be recorded. Results will be expressed in cmH₂O and as a percentage of age- and sex-predicted reference values. Infection control procedures will include disposable, single-use mouthpieces and filters.
Maximal Expiratory Pressure (MEP) | Baseline and Week 8 (Post-Intervention)
  Maximal Expiratory Pressure (MEP) will be assessed using a portable electronic mouth pressure device (Micro Medical Micro RPM, UK). The participant will first perform maximal inspiration, then exhale maximally against an occluded airway for 1-3 seconds. The best of three measurements will be used. Data will be reported in cmH₂O and as a percentage of predicted values based on age and sex. Standard infection control measures with single-use mouthpieces and filters will be followed.
Biceps Brachii Muscle Strength | At baseline and at the end of the 8th week of intervention.
  Quantitative strength of the biceps brachii muscle will be measured using a portable handheld dynamometer (MicroFET2, Hoggan Scientific, USA) with the patient seated in a chair with back support. Both dominant and non-dominant sides will be assessed. The "make test" method will be used, where the assessor holds the device stable while the participant applies maximal force. Three measurements will be taken with 60-second rest intervals, and the mean value will be recorded.
Quadriceps Femoris Muscle Strength | At baseline and at the end of the 8th week of intervention.
  Quantitative strength of the quadriceps femoris muscle will be measured using a portable handheld dynamometer (MicroFET2, Hoggan Scientific, USA) with the patient seated in a chair with back support. Both dominant and non-dominant sides will be assessed. The "make test" method will be used, with three trials taken and 60-second rests in between. The mean of the three measurements will be recorded.
Handgrip Strength | At baseline and at the end of the 8th week of intervention.
  Handgrip strength will be measured using a manual hydraulic dynamometer (Jamar®, California, USA) with the patient seated in a chair with back support. Both dominant and non-dominant hands will be assessed. The "make test" method will be applied, and participants will perform three trials with 60-second rests. The average of the three trials will be recorded.
Sit-Up Test | At baseline and at the end of the 8th week of intervention.
  Core muscle strength will be assessed using the sit-up test. Participants will lie on a mat with knees flexed at 90°, hands behind the head, and feet stabilized. They will be asked to flex the trunk until the inferior angle of the scapula leaves the mat. The number of repetitions completed in 30 seconds will be recorded.
Modified Push-Up Test | At baseline and at the end of the 8th week of intervention.
  Core muscle strength will also be assessed using the modified push-up test. Starting in a prone position with elbows, hands, and knees flexed, participants will be asked to extend their elbows fully and lift the head, shoulders, and trunk off the ground. The number of repetitions completed in 30 seconds will be recorded.
Trunk Flexion Endurance Test | At baseline and at the end of the 8th week of intervention.
  Participants will sit with the trunk supported at 60° flexion, knees bent, and feet flat on the mat. After removing support, they will hold the flexed trunk position as long as possible. Time will be recorded in seconds.
Trunk Extension Endurance Test | At baseline and at the end of the 8th week of intervention.
  Participants will lie prone with the anterior superior iliac spines aligned at the edge of a table. With the upper body unsupported, they will cross their arms and hold the trunk in a horizontal position as long as possible. Time will be recorded in seconds
Right Side Bridge Endurance Test | At baseline and at the end of the 8th week of intervention
  Participants will lie on the right side with feet stacked and the right elbow placed on the mat. They will lift their hips to maintain a straight line from head to feet and hold the position as long as possible. Time will be recorded in seconds.
Left Side Bridge Endurance Test | At baseline and at the end of the 8th week of intervention.
  Participants will lie on the left side with feet stacked and the left elbow placed on the mat. They will lift their hips to maintain a straight line from head to feet and hold the position as long as possible. Time will be recorded in seconds.
Six-Minute Walk Test (6MWT) | At baseline and at the end of the 8th week of intervention.
  Functional capacity will be assessed using the six-minute walk test. Participants will rest for 10 minutes before the test. Heart rate, blood pressure, oxygen saturation, respiratory rate, dyspnea, and fatigue perception will be recorded before and after the test. Dyspnea and fatigue will be assessed with the Modified Borg Scale, and heart rate and oxygen saturation will be measured using a portable pulse oximeter. The test will be conducted in a 30-meter marked corridor, where participants will be asked to walk as far as possible at a fast but comfortable pace for 6 minutes. Rest periods during the test will be recorded with reasons. The total distance walked in meters will be used as the test score.
Static Balance (Romberg Test) | At baseline and at the end of the 8th week of intervention.
  Static balance will be assessed using the TechnoBody PK 252 system with the Romberg test. Participants will stand on the platform in both stable and unstable conditions, with eyes open (30 seconds) and eyes closed (30 seconds). Balance will be evaluated by sway area (mm²) and perimeter (mm).
  Time Frame: At baseline and at the end of the 8th week of intervention.
Dynamic Balance (Limits of Stability Test) | At baseline and at the end of the 8th week of intervention.
  Dynamic balance will be assessed using the TechnoBody PK 252 system with the Limits of Stability Test. Participants will shift their weight to move a cursor toward visual targets appearing in eight directions without lifting their feet. Success rate (%) in reaching the targets will be recorded under both stable and unstable platform conditions.
Diaphragm Thickness | At baseline and at the end of the 8th week of intervention.
  Diaphragm thickness will be assessed using B-mode ultrasound with an 8-15 MHz linear probe placed at the 8th intercostal space in the zone of apposition. Measurements will be taken at end-expiration and at maximal inspiration. The thickening fraction (%) will be calculated as: (inspiratory thickness - expiratory thickness) / expiratory thickness × 100.
Transversus Abdominis Muscle Thickness | At baseline and at the end of the 8th week of intervention.
  Transversus abdominis thickness will be measured with the participant in the supine position using a linear probe placed in the transverse plane at the mid-axillary line above the iliac crest. Measurements will be taken at rest and during the abdominal drawing-in maneuver to activate deep abdominal muscles. The average of three trials will be recorded.
Quadriceps Femoris Muscle Thickness | At baseline and at the end of the 8th week of intervention.
  Thickness of the quadriceps femoris (rectus femoris and vastus intermedius) will be measured by ultrasound with the participant in the supine position and knees fully extended. The probe will be placed at the midpoint of the line between the anterior superior iliac spine and the upper border of the patella. The average of three trials will be recorded for each side.

SECONDARY OUTCOMES:
Physical Activity (Accelerometer Assessment) | At baseline and at the end of the 8th week of intervention.
  Physical activity will be objectively assessed using a triaxial accelerometer (Actigraph wGT3X+). Participants will be instructed to wear the device for 7 consecutive days, removing it only during water-based activities. A minimum of 4 valid days (including 1 weekend day) with at least 10 hours of wear time per day will be required for data inclusion. The device records activity counts, intensity, and energy expenditure across three axes, with vector magnitude calculated. Data will be analyzed using ActiLife6 software. Outcomes will include sedentary time, total physical activity, light physical activity, and moderate-to-vigorous physical activity (MVPA). Compliance with the physical activity guideline of at least 60 minutes of MVPA per day will also be evaluated (yes/no).
Posture Assessment | At baseline and at the end of the 8th week of intervention.
  Posture will be assessed using the validated PostureScreen® Mobile application. Three standardized photographs (anterior, right lateral, and left lateral) will be taken with the smartphone camera using a vertical axis as reference. Anatomical reference points will be marked, and deviations from the midline will be analyzed.
Quality of Life (Leicester Cough Questionnaire - LCQ) | At baseline and at the end of the 8th week of intervention.
  Quality of life will be assessed using the Leicester Cough Questionnaire (LCQ), a 19-item, 7-point Likert-type scale with three subdomains: physical (8 items), psychological (7 items), and social (4 items). Lower scores indicate greater impairment from cough, while higher scores indicate less impact. The Turkish version of the scale has been validated and found reliable.
Patient Satisfaction (Telemedicine Satisfaction Questionnaire - TSQ) | At the end of the 8th week of intervention.
  Patient satisfaction with remote rehabilitation will be assessed using the Telemedicine Satisfaction Questionnaire (TSQ). This validated 14-item scale uses a 5-point Likert format, with total scores ranging from 14 to 70. Higher scores indicate greater satisfaction with telemedicine-based rehabilitation services.
Treatment Adherence (Exercise Diary) | During the 8-week intervention.
  Participants will record their daily exercise participation in a diary throughout the 8-week intervention. Exercise diaries will be used to monitor adherence to the prescribed training program.
Perceived Health Change (Global Rating of Change - GROC) | At the end of the 8th week of intervention.
  Perceived improvement or worsening in health status will be assessed using the Global Rating of Change (GROC) Scale. This 7-point scale ranges from -3 ("much worse") to +3 ("completely recovered"), with higher scores indicating greater perceived improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul,, Istanbul, Turkey (Türkiye)